CLINICAL TRIAL: NCT04837625
Title: A Multicenter Prospective Registration Study of Myasthenic Crisis in China
Brief Title: Study of Myasthenic Crisis in China
Status: Recruiting | Type: Observational
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Chongbo Zhao, Professor, Huashan Hospital
Other Study IDs: MC2020883
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Myasthenia Gravis; Myasthenic Crisis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Myasthenic Crisis Cohort
  Interventions: Other: no interventions

INTERVENTIONS:
Other: no interventions — no interventions

SUMMARY:
This study is a multicenter, prospective, observational research. It will register the basic demographic information, medical history characteristics, clinical features, auxiliary examinations, treatment, outcomes of tracheal intubation/ventilator related events, and clinical outcomes of Myasthenic Crisis patients. The objectives including:

1. Obtain epidemiological data of MC in China;
2. Establish a standardized registration system for MC patients in China;
3. Explore the epidemiology, clinical characteristics, serological characteristics, clinical characteristics of MC, predisposing and predictive factors, extubation process/time, weaning/extubation outcome and predictors of clinical outcome in Chinese MC patients.

ELIGIBILITY:
Inclusion Criteria:

* clinical history and signs of fluctuating weakness and fatigability;
* seropositivity forAChR/MuSKantibodies;
* If negative or the tested antibodies, positive repetitive nerve stimulation(RNS) at low frequency(2-5Hz) is required;
* Crisis: a serious, life-threatening, rapid worsening of MG requiring intubation or noninvasive ventilation to avoid intubation.
* Impending crisis: rapid clinical worsening of MG that, in the opinion of the treating physician, could lead to crisis in the short term (days to weeks) with blood gases suggest hypoxia (oxygen saturation <95%) or elevated carbon dioxide (paco2>50mmHg).

Exclusion Criteria:

* the RNS had over 100% increase after high frequency stimulation or R2 repeats,to differentiate from lambert-Eaton syndrome and congenital MG.
* except when intubation or noninvasive ventilation are employed during routine postoperative management.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be recruited from multiple centers across China.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
MG-ADL of 3 years after off-mechanical ventilation | Sep,2026

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital Fudan University, Shanghai, Shanghai Municipality, China